CLINICAL TRIAL: NCT03872713
Title: Induced Pluripotent Stem Cells for the Development of Novel Drug Therapies for Hepatic and Neurological Morquio Disease
Brief Title: Establishment of Human Cellular Disease Models for Morquio Disease
Acronym: IPSMORQUIO
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: IPSM 09-2018
Record Dates: First submitted 2019-03-06; First posted 2019-03-13 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Morquio Disease
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The skin biopsy will be carried out for patients with a diagnosis of Niemann Pick. The biopsy is performed by the physician by means of punch biopsy (diameter 2-3 mm) under local anesthesia, preferably on the forearm (alternatively: thigh). The biopsy is immediately transferred to sterile cell culture medium and sent by center representative for the quickest possible processing to CENTOGENE's laboratory located in Germany or to professional collaborators being part of the project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establishment of human cellular disease models for Morquio disease for an individualized therapy development having the capacity to address both hepatic and neurologic forms of the disease

DETAILED DESCRIPTION:
The mucopolysaccharidoses are a group of inherited lysosomal storage disorders. Lysosomes function as the primary digestive units within cells. Enzymes within lysosomes break down or digest particular nutrients, such as certain carbohydrates and fats. In individuals with MPS disorders, deficiency or malfunction of specific lysosomal enzymes lead to an abnormal accumulation of certain complex carbohydrates (mucopolysaccharides or glycosaminoglycans) in the arteries, skeleton, eyes, joints, ears, skin and/or teeth. These accumulations may also be found in the respiratory system, liver, spleen, central nervous system, blood, and bone marrow. This accumulation eventually causes progressive damage to cells, tissues, and various organ systems of the body. There are several different types and subtypes of mucopolysaccharidosis. These disorders, with one exception, are inherited as autosomal recessive traits and all vary in their clinical phenotype. Within our clinical trial we focus on MPS type IV.

Morquio syndrome (mucopolysaccharidosis type IV; MPS IV) is a mucopolysaccharide storage disease that exists in two forms (Morquio syndromes A and B) and occurs because of a deficiency of the enzymes N-acetyl-galactosamine-6-sulfatase and beta-galactosidase, respectively. A deficiency of either enzyme leads to the accumulation of mucopolysaccharides in the body, abnormal skeletal development, and additional symptoms. In most cases, individuals with Morquio syndrome have normal intelligence. The clinical features of MPS IV-B are less severe than those associated with MPS IV-A. Symptoms may include growth retardation, a prominent lower face, an abnormally short neck, knees that are abnormally close together (knock knees or genu valgum), flat feet, abnormal sideways and front-to-back or side-to-side curvature of the spine (kyphoscoliosis), abnormal development of the growing ends of the long bones (epiphyses) resulting in dwarfism, and/or a prominent breast bone (pectus carinatum) as well as bell shaped chest. Though the CNS and peripheral nerves are primarily not affected the bone defects may result in neurological symptoms such as spinal cord compression. Hearing loss, weakness of the legs, and/or additional abnormalities may also occur.

The goal of the study is to prepare a cell culture from patients affected with Morquio disease in order to identify novel pathways and proteins involved in disease progression that allow for an earlier diagnosis (i.e. before symptom onset) and that are suitable targets for an individualized therapeutic approach able to address not only the hepatic form, but also the neurologic form of the disease, which is less responsive to the current therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures
* Patients of both genders older than 12 months
* Patient has a diagnosis of Morquio disease

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures
* Patient is younger than 12 months
* Patient has no diagnosis of Morquio disease

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient has a diagnosis of Morquio disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Reprogramming patient-derived fibroblasts into induced pluripotent stem cells | 24 months
  The aim of this study is to generate patient-specific induced pluripotent stem cells and then differentiate them into chondrocytes to study the accumulation of keratin sulfate (KS) and chondroitin-6-sulfate (C6S), and possible mechanism to reduce the accumulated substances and modulate the defective enzyme

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, Prof. Dr., Principal Investigator — CENTOGENE GmbH Rostock
Locations (1):
- Childrens Hospital and Institute of Child Health, Ferozepur Road, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided